CLINICAL TRIAL: NCT03946852
Title: Abdominal Regional Perfusion in Donation After Cardiac Death for Multi-Organ Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Ephraim Tang, Clinical Fellow, Multi-Organ Abdominal Transplant, London Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113712
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Liver Transplant; Complications; Ischemia Reperfusion Injury; Cirrhosis; Liver Cancer; Liver Metastases; End Stage Liver Disease
Keywords: abdominal regional perfusion; Donation after Cardiac Death; Liver Transplantation; Ischemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury; Fibrosis; Liver Neoplasms; End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARP arm (Experimental): Patients will receive DCD after therapy after the abdominal reperfusion protocol.
  Interventions: Device: Abdominal Regional Perfusion

INTERVENTIONS:
Device: Abdominal Regional Perfusion — Abdominal Regional Perfusion

SUMMARY:
The main purpose of this study is to increase the pool of organs available for donation by performing ARP to recondition donation after cardiac death (DCD) organs prior to transplantation. We will compare the outcomes of our ARP DCD liver transplants with historical data to determine the efficacy of this treatment compared to transplantation with standard DCD and donation after brain death (DBD) organs. We will also analyze biological samples from donors and recipients and compare them with outcome data in an effort to determine if any biological markers are able to predict the quality/success of the grafts.

DETAILED DESCRIPTION:
Liver Transplantation and Limitations of DCD Transplantation:

Liver transplantation (LT) is the sole curative therapy for end stage liver disease and has emerged as the treatment of choice for hepatocellular carcinoma. Recent evidence has also demonstrated efficacy in a growing number of malignancies including intra/extra-hepatic cholangiocarcinoma, metastatic neuro-endocrine tumors, and colorectal liver metastases. Despite these advantages, LT is limited by the availability of suitable donor organs resulting in lengthened LT waitlist times. However, during this waiting period patients may deteriorate making them ineligible for LT. In the US, 16,000 patients are listed for LT, and approximately 2000 die annually while waiting for suitable organs. In 2017, over 500 Canadians were on a waiting list for LT and nearly 200 died or withdrew from the transplant list while waiting. Additionally, while LT secondary to hepatitis C is declining, nonalcoholic steatohepatitis, alcoholic liver disease and transplant oncology indications are growing, increasing the overall demand for liver transplant.

One strategy to expand the donor pool has been to optimize utilization of organs from donation after cardiac death (DCD). While outcomes of DCD kidney, pancreas and lung transplants show similar patient and graft survival to donation after brain death (DBD) transplants, DCD livers have worse patient and graft survival, higher complications, and costs, along with worse quality of life. DCD liver grafts have twice the rate of early complications including primary non-function (PNF) and early allograft dysfunction (EAD). EAD is a transient condition with the potential for graft function recovery whereas PNF is a more severe complication leading to graft failure requiring emergency re-transplantation. In the long term, the use of DCD liver allografts is associated with a 10 fold increase in biliary complications, typically resulting in graft loss or death. Moreover, there is a high cost associated with complications and readmissions following LT, which can be upwards of $50,000 per patient. Studies investigating factors contributing to these costs have revealed that DCD allografts had the greatest impact on transplant costs. Consequently, initial enthusiasm for the use of DCD livers for LT has waned such that utilization is restricted to only ideal DCD livers from younger donors with short warm and cold ischemia times. Developing methodologies to reduce the complications associated with DCD organs and improve overall outcomes would have an immense impact on the lives of transplant patients while concurrently reducing costs on the healthcare system.

Abdominal Regional Perfusion and Limitations of Normothermic Machine Perfusion:

Conventional DCD recovery utilizes a rapid recovery technique which flushes abdominal organs with cold preservation solution to slow cellular metabolism and evacuate blood/clots to preserve the integrity of the microvasculature. This is preceded by the agonal phase between withdrawal of life support and cessation of cardiac function. During this period, abdominal organs are subject to warm ischemia resulting in accumulation of toxic metabolites, depletion of intracellular energy and anti-oxidant stores, leading to exacerbation of ischemia reperfusion at the time of implantation.

Abdominal Regional Perfusion (ARP) is a technique that has been developed to recondition DCD organs prior to transplantation through the perfusion of abdominal organs in-situ with re-oxygenated blood. This process reverses the effects of ischemia and hypoxia by restoring cellular energy stores and reducing oxygen free-radicals. Additionally, this period of restored abdominal perfusion also allows for functional evaluation of organ viability prior to graft use through measurement of donor serum/bile biochemistry throughout the perfusion process, thereby maximizing the yield of high quality grafts and avoiding the use of grafts that have impaired function.

In the few studies published to date, ARP has demonstrated a decrease in biliary complications by 86%, a decrease in ischemic cholangiopathy rates from 27% to 0% and a drop in EAD from 32% to 12%. Most importantly, graft loss at 30 days was only 2% in ARP compared with 12% in conventional DCD LT. Emerging evidence suggests that with ARP, transplants performed using DCD organs can result in outcomes similar to conventional DBD donors. In addition, other investigators have successfully used ARP to further expand the DCD donor pool by including donors beyond the traditional age limit of 50 years to patients greater than 75. This approach has the potential to dramatically increase the donor pool and has even been demonstrated to improve the quality of other organs used for transplant including kidney and heart transplantation.

Although normothermic machine perfusion (NMP) systems have demonstrated non-inferiority compared to static cold storage in LT by dropping perfusate lactate, improving intraoperative mean arterial pressure, reducing vasopressor requirements and reducing blood product transfusions, the majority (80%) of these donor livers were procured from DBD donors in which static cold storage continues to be the standard of care based upon three decades of favorable outcomes. There remains a paucity of data demonstrating the benefit of NMP in the setting of expanded criteria livers from donors with advanced age, steatosis, and DCD livers where ARP has been of proven benefit. In addition, ARP may also be advantageous due to its in-situ nature with preservation of the neurohormonal axis and communication with other abdominal organs. Few clinical studies have investigated the role of measurable variables in predicting ARP-DCD transplant outcomes; however, some correlation has been found between the effects of lactate levels, transaminase levels and the level of fibrosis on donor organ function. To address these unknowns, an additional goal of this study will be to identify possible mediators for the improved outcomes with abdominal-regional perfusion, and evaluate the utility of biomarkers to predict graft function.

ELIGIBILITY:
Recipient Criteria:

Inclusion Criteria- Indications for Liver transplant include decompensated Cirrhosis of any etiology Model for End-Stage Liver Disease (MELD) score > 15 with no contraindications to liver transplant as per conventional clinical practice.

Acute or fulminant liver failure Advanced malignancy such as HCC, cholangiocarcinoma, neuroendocrine tumor, or other cancer meeting criteria for listing and exception points as per current clinical guidelines.

Exclusion Criteria-

* Inadequate social support for liver transplant
* Non-compliance with alcohol or narcotic cessation
* Evidence of uncontrolled infection
* Other untreated malignancy aside from those listed above
* Physiologic evidence of frailty based on timed up and go, grip strength, 6 minute walk test, and cognitive testing.

Donor Criteria:

DCD donors offered via TGLN will be considered for assessment via abdominal regional perfusion based on the following parameters. These are in keeping with current criteria for abdominal organ donors.

* Age: Up to 70 years of age within the initial evaluation period, with plans to expand to 75 y/o if initial results are favourable.
* BMI: Donor BMI must be less than 30 for consideration
* DCD donation criteria: Conventional criteria for DCD donation must be met, including no expectation for viable recovery, without meeting criteria for brain death, and expressed desire by family for organ donation.
* Comorbidity: In the opinion of the on-call transplant surgeon, there should not be excessive comorbidity to exclude organ donation
* Active infection: There should be no untreated infection.
* Malignancy: Donors should have no evidence of active malignancy, or in the case of a treated malignancy there should be sufficient interval to rule out recurrence. In select cases, donors with tumors known to be indolent may be considered on a case by case basis.

Liver transplant release Criteria:

One of the major advantages of ARP beyond reconditioning the organ prior to cold storage and transplant, is an opportunity to assess graft function in-situ prior to transplant. The existing literature supports the use of multiple readily available laboratory tests to evaluate graft function prior to transplant. Donor labs will be drawn every 30 minutes from the perfusion circuit to evaluate organ function.

* Transaminase: Initial transaminases (AST and ALT) drawn at the start of perfusion must be less than 4 times the upper limit of normal and stay below this threshold throughout the reperfusion process to be considered for use with an absolute cut-off of 500
* Lactate: Grafts will only be used if lactate levels do not rise during perfusion, ideal organs will have a decrease in serum lactate levels by 1.11 mmol/L per hour
* Macroscopic appearance: On clinical evaluation, there should be no evidence of fibrosis or cirrhosis and organs should not have a macroscopically steatotic appearance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary non-function | 1 week
  Graft failure requiring re-transplantion
Early allograft dysfunction | 1 week
  Transient non-functioning of the liver transplant but with usual recovery to full functioning liver
Ischemic Cholangiopathy | 1 week to 12 months post transplant
  Non-anastomotic biliary stricture without other identifiable etiology

SECONDARY OUTCOMES:
Overall patient survival | 1 and 5 years
  Patient Mortality at any time post transplant
Graft survival | 5 years
  Need for retransplant secondary to graft failure of any cause, or death

OTHER OUTCOMES:
Biliary anastomotic stricture | 1 year
  Imaging or biochemical evidence of anastomotic stricture requiring intervention
Biliary Anastomotic leak | 30 days
  Imaging or endoscopic evidence of bile leak requiring antibiotics or percutaneous drainage
Length of ICU stay | 30 days
  Duration of post-operative stay in ICU
Overall Length of stay | 30 days
  Overall duration of stay in hospital post-transplant
Re-operation rate | 30 days
  Frequency of return to the operating room for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim S Tang, MD, MSc, Principal Investigator — Clinical Fellow; Anton I Skaro, MD, PhD, Principal Investigator — Transplant Surgeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Hessheimer AJ, Garcia-Valdecasas JC, Fondevila C. Abdominal regional in-situ perfusion in donation after circulatory determination of death donors. Curr Opin Organ Transplant. 2016 Jun;21(3):322-8. doi: 10.1097/MOT.0000000000000315. PMID 27050485
- [Background] Watson CJE, Hunt F, Messer S, Currie I, Large S, Sutherland A, Crick K, Wigmore SJ, Fear C, Cornateanu S, Randle LV, Terrace JD, Upponi S, Taylor R, Allen E, Butler AJ, Oniscu GC. In situ normothermic perfusion of livers in controlled circulatory death donation may prevent ischemic cholangiopathy and improve graft survival. Am J Transplant. 2019 Jun;19(6):1745-1758. doi: 10.1111/ajt.15241. Epub 2019 Feb 1. PMID 30589499
- [Background] Ruiz P, Gastaca M, Bustamante FJ, Ventoso A, Palomares I, Prieto M, Fernandez JR, Salvador P, Pijoan JI, Valdivieso A. Favorable Outcomes After Liver Transplantation With Normothermic Regional Perfusion From Donors After Circulatory Death: A Single-center Experience. Transplantation. 2019 May;103(5):938-943. doi: 10.1097/TP.0000000000002391. PMID 30063694
- [Background] Jay CL, Lyuksemburg V, Ladner DP, Wang E, Caicedo JC, Holl JL, Abecassis MM, Skaro AI. Ischemic cholangiopathy after controlled donation after cardiac death liver transplantation: a meta-analysis. Ann Surg. 2011 Feb;253(2):259-64. doi: 10.1097/SLA.0b013e318204e658. PMID 21245668